CLINICAL TRIAL: NCT05008419
Title: Remediating Narrative Discourse Impairments in Veterans With TBI: Initial Treatment Development
Brief Title: Narrative Discourse Treatment Development
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3494-W; 1IK2RX003494-01A2 (NIH)
Record Dates: First submitted 2021-08-09; First posted 2021-08-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Traumatic Brain Injury; Neurogenic Communication Disorders
Keywords: traumatic brain injury; neurogenic communication disorders; pragmatic communication disorders
MeSH Terms: conditions — Brain Injuries, Traumatic; Communication Disorders; Social Communication Disorder

STUDY DESIGN:
Intervention Model Description: 40 participants with TBI will be randomized to receive the discourse treatment with a telehealth component or Treatment as Usual (TAU).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Discourse Treatment (Experimental): Biweekly discourse treatment sessions.
  Interventions: Behavioral: Narrative discourse treatment
- Treatment as Usual (No Intervention): No treatment. Participants will engage in their usual care.

INTERVENTIONS:
Behavioral: Narrative discourse treatment — The protocol will incorporate elements from prior treatment studies that showed some promise: 1) hierarchical training, 2) variety of discourse stimuli, 3) development of skills and strategies for discourse processing, 4) structured training prompts, 5) meta-cognitive and meta-linguistic strategies, and 6) integration of learning principles. Novel treatment elements will include: 1) targeting both story content and story organization, 2) use of a discourse model to guide treatment, and 3) functional communication training. Treatment will be delivered twice a week over 8 weeks. There will be four treatment phases: education, story organization, story content, and integration of story organization and content.
  Arms: Discourse Treatment

SUMMARY:
Discourse impairments are breakdowns in meaningful communication beyond the level of single sentences and have a functional impact on the lives of Veterans with TBI, disrupting return to work, communication re integration, socialization, and quality of life. The few prior attempts to treat discourse impairments have been small case studies and resulted in no change or limited gains. The proposed study evaluates the feasibility of a novel narrative discourse treatment that builds upon these prior attempts by addressing breakdowns in both story content and story organization using a theoretically-driven approach. If feasible, as demonstrated by tolerability and acceptability to participants, and later shown to be effective, the proposed discourse treatment has the potential to improve daily communication, which provides a gateway for Veterans with TBI to increase meaningful participation and improve functioning in major life domains.

DETAILED DESCRIPTION:
Discourse intervention in TBI is a nascent area of research, and, to date, there have been only a few studies that have attempted to improve discourse ability in TBI. These prior attempts have been small case studies, produced no change or limited gains, and did not include Veterans with TBI. The proposed project is an early stage discourse treatment development study that will evaluate the feasibility of a novel narrative discourse treatment protocol that builds upon these prior attempts with an all-Veteran participant sample. The first part of the study will consist of initial manual development for the discourse treatment protocol and refinement.

The second part will involve a treatment feasibility trial to obtain information regarding the tolerability, acceptability, and fidelity of the proposed discourse treatment and preliminary data on treatment delivery and assessment methods as well as preliminary information about treatment effects. Forty participants will be randomized to either the discourse treatment group or Treatment as Usual control. Assessments will be conducted at baseline, post-treatment, and at 1-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Veteran with diagnosis of TBI with mild to moderate functional cognitive impairments
* Self-report of communication difficulty following TBI that interferes with activities
* Can identify a significant other (e.g., spouse, family member, friend) who is able and willing to serve as an informant, who will verify discourse ability pre- and post-treatment

  * The informant must be an individual with whom the participant engages in weekly social communication
* Adequate hearing and visual acuity to participate in study procedures
* Those who are willing and able to participate in telehealth sessions must have appropriate equipment and access

  * e.g., smartphone, tablet, computer with camera, internet access
* Stable housing

  * Participants must have a safe, private and quiet environment in their home to engage in telehealth sessions
* English as a primary language

Exclusion Criteria:

* Penetrating head injury
* History of or current developmental disability (e.g., dyslexia), psychotic disorder, neurological illness

  * e.g., stroke, dementia, Parkinson's disease), aphasia or auditory processing disorder (APD)
* Current (past 30 days) diagnosis of alcohol or substance abuse

  * An exception will be made for marijuana as a number of Veterans use marijuana occasionally to manage ailments, such as pain and PTSD
  * Marijuana use must not occur regularly or interfere with daily functioning
  * Inclusion of Veterans using marijuana aligns with the VA's position that Veterans will not be denied VA benefits because of marijuana use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Tolerability of treatment as measured by rates of attendance for all aspects of treatment | 2 months
  Rates of attendance for all aspects of treatment, calculated as the number of treatment sessions attended across all treatment phases divided by total number of treatment sessions.
Feasibility of treatment as measured by dropout rate in the treatment condition | 2 months
  Dropout rate in the treatment condition will be calculated as the number of participants who do not complete treatment over total number of participants
Acceptability of treatment as measured by a treatment satisfaction survey | 2 months
  Percentage of participants who rate satisfaction with the treatment based on Likert-type survey (e.g., endorse "satisfied" or "very satisfied")

CONTACTS AND LOCATIONS:
Overall Officials: Karen Le, PhD, Principal Investigator — VA Connecticut Healthcare System West Haven Campus, West Haven, CT
Locations (1):
- VA Connecticut Healthcare System West Haven Campus, West Haven, CT, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Final data sets underlying all publications resulting from the research may be shared as per access criteria delineated below.
Time Frame: 6 months after publication
Access Criteria: De-identified data sets may be shared with other investigators, upon written request, under a data use agreement prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset. The data sharing agreement will also restrict redistribution to third parties and proper acknowledgment of the data source. These data sets will be shared per guidelines provided by the VA Connecticut Healthcare System (VACHS) Information Security Officer.

DOCUMENTS (1):
  • Informed Consent Form (2024-02-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT05008419/ICF_000.pdf